CLINICAL TRIAL: NCT03824418
Title: The Clinical Value of Chromoendoscopy as Surveillance Strategy for Dysplasia Detection in Ulcerative Colitis: an Observational Follow-up Study
Brief Title: The Clinical Value of Chromoendoscopy as Surveillance Strategy for Dysplasia Detection in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 00001
Record Dates: First submitted 2018-03-09; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis; Chromoendoscopy
Keywords: Surveillance; Chromoendoscopy; Dysplasia; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chromoendoscopy follow-up
  Interventions: Procedure: Surveillance colonoscopy with chromoendoscopy
- Autofluorescence follow-up
  Interventions: Procedure: Surveillance colonoscopy with chromoendoscopy

INTERVENTIONS:
Procedure: Surveillance colonoscopy with chromoendoscopy — Surveillance colonoscopy with chromoendoscopy

SUMMARY:
A recent multicentre randomised controlled trial compared autofluorescence imaging (AFI) with CE for dysplasia detection in colonoscopy surveillance of patients with longstanding UC (FIND-UC). In this study, CE detected significantly more dysplastic lesions per patient compared with AFI. It is unclear whether this increased dysplasia detection also translates to a reduction of dysplasia at follow-up colonoscopy. The aim of this pre-specified study is therefore to prospectively determine whether there is a difference in dysplasia detection at follow-up colonoscopy between UC patients who were randomized to AFI or CE at index colonoscopy for the FIND-UC trial.

ELIGIBILITY:
Patients are eligible for inclusion in this study when they meet the following criteria:

Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

- Patients that where included in the previous FIND-UC trial

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Patients who not receive their surveillance colonoscopy with CE
* Patients who not undergo their surveillance colonoscopy within 3 months of the surveillance recommendations

Withdrawal of individual subjects

A patient will be excluded from the study if any of the following events occur:

* Withdrawal of informed consent
* The patient requests to be discontinued from the study
* The bowel preparation is scored as Boston Bowel Preparation Scale <6
* Incomplete colonoscopy because the endoscopist is unable to intubate the cecum during the colonoscopy
* The Mayo-score > 1 in at least in one of the bowel segments

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of the FIND-UC trial that undergo a follow surveillance colonoscopy
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
the proportion of patients in which at least one histological proven dysplastic lesions was detected at follow-up colonoscopy. | during surveillance colonoscopy
  the proportion of patients in which at least one histological proven dysplastic lesions was detected at follow-up colonoscopy.

SECONDARY OUTCOMES:
The proportion of patients in which at least one histological proven neoplastic lesion was detected | during surveillance colonoscopy
  The proportion of patients in which at least one histological proven neoplastic lesion was detected
The mean number of histological proven neoplastic lesions per patient | during surveillance colonoscopy
  The mean number of histological proven neoplastic lesions per patient
The proportion of patients in which at least one histological proven sessile serrated lesion was detected | during surveillance colonoscopy
  The proportion of patients in which at least one histological proven sessile serrated lesion was detected
The mean number of histological proven sessile serrated lesions per patient | during surveillance colonoscopy
  The mean number of histological proven sessile serrated lesions per patient
Description of dysplasia detected at follow-up colonoscopy (colonic segment, location with respect to a resection scar if visible), or in the resection specimen after proctocolectomy. The proportion of lesions defined as new/missed and recurrent lesion | during surveillance colonoscopy
  Description of dysplasia detected at follow-up colonoscopy (colonic segment, location with respect to a resection scar if visible), or in the resection specimen after proctocolectomy. The proportion of lesions defined as new/missed and recurrent lesions detected during surveillance colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol